CLINICAL TRIAL: NCT01781429
Title: Phase I Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of BVD-523 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVD-523-01; BVD-523-01 (Other: BioMed Valley Discoveries, Inc.)
Record Dates: First submitted 2013-01-28; First posted 2013-02-01 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — ulixertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BVD-523 (Experimental)
  Interventions: Drug: BVD-523

INTERVENTIONS:
Drug: BVD-523 — Oral, multiple escalating doses, twice daily, for 21 days in each treatment cycle

SUMMARY:
This open-label, multi-center Phase 1/2 study will assess the safety, pharmacokinetics, and pharmacodynamics of escalating doses of BVD-523 in patients with advanced malignancies. The study also seeks to demonstrate target modulation and early signs of clinical response in select patient populations.

DETAILED DESCRIPTION:
The study is being performed to assess the safety and tolerability of BVD-523

In Part 1 of the study, an accelerated dose escalation plan will be used to establish dose limiting toxicities, maximum tolerated dose, and the recommended Phase 2 dose.

In Part 2 of the study, additional patients with particular tumor types and/or cancers harboring specific genetic mutations will be recruited for treatment at the Recommended Phase 2 Dose. Patients may also be assessed pharmacodynamic measures in healthy or malignant tissues, using biomarker assays for phosphorylation, cytotoxic or cytostatic measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or advanced-stage malignant tumor. Patients may have received up to 2 prior lines of chemotherapy for their metastatic disease
* ECOG score of 0 or 1
* Predicted life expectancy of ≥ 3 months
* Adequate bone marrow, liver and renal function renal function
* Adequate cardiac function
* For women: Negative pregnancy test for females of child-bearing potential; must be surgically sterile, postmenopausal, or compliant with a contraceptive regimen during and for 3 months after the treatment period
* For men: Must be surgically sterile, or compliant with a contraceptive regimen during and for 3 months after the treatment period
* For Part 2 of the Study only, patients must have measurable disease by RECIST 1.1 and be in one of the the groups below. Patients in groups 1, 2, 4, 5 and 6 may not have been previously treated with BRAF and/or MEK inhibitors

  * Group 1: Patients with BRAF mutated cancer, except those with colorectal or non-small cell lung cancers
  * Group 2: Patients with BRAF mutated colorectal cancer
  * Group 3: Patients with BRAF mutated melanoma who have progressed on, or are refractory to BRAF and/or MEK inhibitors
  * Group 4: Patients with NRAS mutated melanoma
  * Group 5: Patients with MEK mutated cancer
  * Group 6: Patients with BRAF mutated non-small cell lung cancer
  * Group 7: Patients with ERK mutated cancer

Exclusion Criteria:

* Gastrointestinal condition which could impair absorption of study medication
* Uncontrolled or severe intercurrent medical condition
* Known uncontrolled brain metastases. Stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants
* Any cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc.) within 28 days or 5 half-lives, whichever is shorter
* Major surgery within 4 weeks prior to first dose
* Any use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of BVD-523.
* Pregnant or breast-feeding women
* Any evidence of serious active infections
* Any important medical illness or abnormal laboratory finding that would increase the risk of participating in this study
* A history or current evidence/risk of retinal vein occlusion or central serous retinopathy
* Concurrent therapy with any other investigational agent
* Concomitant malignancies or previous malignancies with less than 2 years disease-free interval at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UCLA Med-Hematology & Oncology, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists and Research Group (Sarah Cannon Research Institute), Sarasota, Florida
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute Hospital at Vanderbilt, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT M.D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Wu J, Liu D, Offin M, Lezcano C, Torrisi JM, Brownstein S, Hyman DM, Gounder MM, Abida W, Drilon A, Harding JJ, Sullivan RJ, Janku F, Welsch D, Varterasian M, Groover A, Li BT, Lacouture ME. Characterization and management of ERK inhibitor associated dermatologic adverse events: analysis from a nonrandomized trial of ulixertinib for advanced cancers. Invest New Drugs. 2021 Jun;39(3):785-795. doi: 10.1007/s10637-020-01035-9. Epub 2021 Jan 3. PMID 33389388
- [Derived] Mendzelevski B, Ferber G, Janku F, Li BT, Sullivan RJ, Welsch D, Chi W, Jackson J, Weng O, Sager PT. Effect of ulixertinib, a novel ERK1/2 inhibitor, on the QT/QTc interval in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2018 Jun;81(6):1129-1141. doi: 10.1007/s00280-018-3564-1. Epub 2018 Mar 30. PMID 29603015
- [Derived] Germann UA, Furey BF, Markland W, Hoover RR, Aronov AM, Roix JJ, Hale M, Boucher DM, Sorrell DA, Martinez-Botella G, Fitzgibbon M, Shapiro P, Wick MJ, Samadani R, Meshaw K, Groover A, DeCrescenzo G, Namchuk M, Emery CM, Saha S, Welsch DJ. Targeting the MAPK Signaling Pathway in Cancer: Promising Preclinical Activity with the Novel Selective ERK1/2 Inhibitor BVD-523 (Ulixertinib). Mol Cancer Ther. 2017 Nov;16(11):2351-2363. doi: 10.1158/1535-7163.MCT-17-0456. Epub 2017 Sep 22. PMID 28939558

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-escalation 10mg b.i.d. Cohort: Patients received 10mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 20mg b.i.d. Cohort: Patients received 20mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 40mg b.i.d. Cohort: Patients received 40mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 75mg b.i.d. Cohort: Patients received 75mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 150mg b.i.d. Cohort: Patients received 150mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 300mg b.i.d. Cohort: Patients received 300mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 600mg b.i.d. Cohort: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 750mg b.i.d. Cohort: Patients received 750mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Dose-escalation 900mg b.i.d. Cohort: Patients received 900mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 3 weeks.
- Cohort-expansion Group 1: Patients with BRAF mutated cancer, except those with colorectal or non-small cell lung cancers, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 2: Patients with BRAF mutated colorectal cancer, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 3: Patients with BRAF mutated melanoma who had progressed or were refractory to BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 4: Patients with NRAS mutated melanoma, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 5: Patients with MEK mutated cancer, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 6: Patients with BRAF mutated non-small cell lung cancer, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
- Cohort-expansion Group 7: Patients with ERK mutated cancer, not previously treated with BRAF and/or MEK inhibitors. Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
Period: Overall Study
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort | Cohort-expansion Group 1 | Cohort-expansion Group 2 | Cohort-expansion Group 3 | Cohort-expansion Group 4 | Cohort-expansion Group 5 | Cohort-expansion Group 6 | Cohort-expansion Group 7
Started | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 24 | 18 | 21 | 22 | 8 | 16 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 24 | 18 | 21 | 22 | 8 | 16 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 5 | 2 | 3 | 0
Not completed — Disease Progression | 1 | 0 | 1 | 1 | 1 | 4 | 7 | 4 | 6 | 15 | 15 | 15 | 15 | 4 | 11 | 0
Not completed — Unacceptable Toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Patient Condition Changed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Other - as entered by PI in eCRF | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Not completed — Enrolled, but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient from Cohort-expansion group 2 was enrolled, but not treated. Therefore, they were not included in the baseline characteristics or study results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort | Cohort-expansion Group 1 | Cohort-expansion Group 2 | Cohort-expansion Group 3 | Cohort-expansion Group 4 | Cohort-expansion Group 5 | Cohort-expansion Group 6 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 24 | 17 | 21 | 22 | 8 | 16 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 3 | 6 | 12 | 7 | 16 | 11 | 6 | 6 | 72
  >=65 years | 1 | 0 | 0 | 1 | 1 | 4 | 4 | 1 | 1 | 12 | 10 | 5 | 11 | 2 | 10 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 5 | 8 | 7 | 9 | 5 | 1 | 9 | 52
  Male | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 2 | 16 | 10 | 12 | 17 | 7 | 7 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 19 | 15 | 21 | 16 | 8 | 15 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 3 | 0 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 6
  White | 1 | 1 | 1 | 1 | 1 | 3 | 7 | 4 | 5 | 19 | 15 | 20 | 18 | 6 | 15 | 117
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 24 | 17 | 21 | 22 | 8 | 16 | 135

OUTCOME MEASURES:

1. Primary Outcome: Determination of Recommended Phase 2 Dose (RP2D) of BVD-523 by Dose-limiting Toxicities (DLT).
Description: DLT is defined as any BVD-523 related toxicity in the first 21 days of treatment that results in:
  1. ≥Grade 4 hematologic toxicity for >1 day;
  2. Grade 3 hematologic toxicity with complications e.g., thrombocytopenia with bleeding;
  3. ≥Grade 3 non-hematologic toxicity, except untreated nausea, vomiting, constipation, pain and rash (these become DLTs if the adverse event (AE) persists despite adequate treatment), a doubling of aspartate transaminase (AST)/alanine transaminase (ALT) in patients with grade 2 ALT/AST at baseline;
  4. A treatment interruption exceeding 5 days (or an interruption exceeding 7 days for rash, despite adequate treatment) in Cycle 1 (or inability to begin Cycle 2 for > 7 days) due to BVD-523-related toxicity.
Time Frame: As indicated by safety and tolerability during study conduct; ~42 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7
Participants
  Any DLT: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  Any DLT: No | 1 | 1 | 1 | 1 | 1 | 4 | 6 | 2 | 5
  Grade 3 Hematologic Toxicity with Complications: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Grade 3 Hematologic Toxicity with Complications: No | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 3 | 5
  ≥Grade 3 Non-Hematologic Toxicity: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
  ≥Grade 3 Non-Hematologic Toxicity: No | 1 | 1 | 1 | 1 | 1 | 4 | 6 | 2 | 5

2. Secondary Outcome: Characterization of the Time Versus Plasma Concentration Profiles of BVD-523 and Selected Metabolites.
Description: Data provided is for BVD-523.
Time Frame: Samples will be collected on day 1 and day 15 of Cycle 1
Population: Day 1 - Dose-escalation 10mg b.i.d. patient was not calculable. Cohort-expansion numbers do not include those patients that were dose reduced and/or were not at a steady state with 600mg b.i.d. for the Day 15 draw.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort | Cohort-expansion Group 1 | Cohort-expansion Group 2 | Cohort-expansion Group 3 | Cohort-expansion Group 4 | Cohort-expansion Group 5 | Cohort-expansion Group 6
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 24 | 18 | 21 | 22 | 8 | 16
ng/mL
  Cmax Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 23 | 17 | 19 | 20 | 8 | 16
  Cmax Day 1 | NA — Day 1 - Dose-escalation 10mg b.i.d. patient was not calculable. | 14.9 | 100 | 133 | 216 | 765 (234) | 1110 (589) | 1450 (539) | 1430 (1010) | 1180 (501) | 1260 (474) | 1190 (467) | 1230 (840) | 1140 (423) | 1560 (885)
  Cmax Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 7 | 3 | 3 | 17 | 12 | 11 | 15 | 4 | 12
  Cmax Day 15 | 45.7 | 15.8 | 191 | 326 | 459 | 586 (257) | 3090 (1570) | 2290 (1790) | 1730 (401) | 2440 (900) | 1890 (953) | 2340 (962) | 1890 (1060) | 2050 (1570) | 2680 (1520)

3. Secondary Outcome: Clinical Evidence of Tumor Response Assessed by Physical or Radiological Exam.
Description: At enrollment, all study patients had metastatic or advanced-stage malignant tumor for which no curative therapy was known to exist. Patients entering Part 2 additionally had to have measurable disease by RECIST version 1.1. Data shown is best response.
Time Frame: Patients will be evaluated at baseline & at periodic follow-up visits through the time their participation in the study is completion. The best responses presented occurred at different time points for each patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort | Cohort-expansion Group 1 | Cohort-expansion Group 2 | Cohort-expansion Group 3 | Cohort-expansion Group 4 | Cohort-expansion Group 5 | Cohort-expansion Group 6
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 4 | 7 | 4 | 7 | 22 | 13 | 15 | 19 | 5 | 14
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 0 | 1 | 3 | 0 | 3
  Stable Disease | 1 | 1 | 0 | 1 | 1 | 2 | 5 | 0 | 4 | 14 | 8 | 6 | 7 | 2 | 9
  Progressive Disease | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 2 | 4 | 5 | 8 | 9 | 3 | 2

4. Other Pre Specified Outcome: Pharmacodynamic (PD) Response Measured as Percentage Enzyme Inhibition of RSK1 Ser 380 (pRSK)
Description: RSK1, a member of the RSK serine/threonine kinase family, is a direct substrate of the MAP Kinases ERK1 & ERK2. RSK1 and ERK1/2 form an inactive complex in unstimulated cells. Upon activation of the mitogenic pathway, ERK1/2 phosphorylates Thr573, Thr359 and Ser363 on RSK1. Thr573 resides in the activation loop of the carboxy terminal kinase domain of RSK1 and once phosphorylated, enables RSK1 to autophosphorylate Ser380. Phosphorylation of Ser380 on RSK1 can therefore be used as a target biomarker for ERK1 and ERK2 activity. BVD-523 inhibits the activity of ERK. In this study, phosphorylation of RSK1 Ser 380 (pRSK) was used as a target biomarker for assessment of ERK inhibition by BVD-523 in human whole blood samples.
Time Frame: Patients will be evaluated at baseline and on ~day 15 of Cycle 1
Population: The protocol was amended to stop collecting PD samples unless the patient consented to a tumor biopsy. Therefore, some patients did not have PD samples collected or did not consent to optional research tests involving collection of tumor tissue and blood/plasma samples.
Measure: Mean (Standard Deviation); unit: Enzyme inhibition (%)
Arm/Group | Cohort-expansion Group 1 | Cohort-expansion Group 2 | Cohort-expansion Group 3 | Cohort-expansion Group 4 | Cohort-expansion Group 5 | Cohort-expansion Group 6
Number analyzed (Participants) | 24 | 17 | 21 | 22 | 8 | 16
Enzyme inhibition (%)
  Cycle 1, Day 1; pre-dose: number analyzed (Participants) | 18 | 6 | 18 | 14 | 6 | 10
  Cycle 1, Day 1; pre-dose | 0.000 (0) | 0.000 (0) | 0.000 (0) | 0.000 (0) | 0.000 (0) | 0.000 (0)
  Cycle 1, Day 1; 4 hours post-dose: number analyzed (Participants) | 18 | 6 | 15 | 14 | 4 | 9
  Cycle 1, Day 1; 4 hours post-dose | 82.162 (27.3012) | 69.989 (36.9362) | 87.563 (26.8634) | 96.868 (5.8054) | 93.910 (12.1800) | 80.214 (28.9393)
  Cycle 1, Day 15; pre-dose: number analyzed (Participants) | 16 | 3 | 11 | 11 | 3 | 7
  Cycle 1, Day 15; pre-dose | 94.607 (9.9291) | 66.667 (57.7350) | 78.679 (37.6286) | 91.955 (21.5915) | 89.050 (18.9660) | 99.447 (1.4627)
  Cycle 1, Day 15; 4 hours post-dose: number analyzed (Participants) | 16 | 4 | 10 | 10 | 3 | 8
  Cycle 1, Day 15; 4 hours post-dose | 91.419 (13.9282) | 56.554 (51.2962) | 87.624 (26.0916) | 98.902 (3.4722) | 92.640 (12.7479) | 85.329 (27.2781)

ADVERSE EVENTS:
Time Frame: The reporting period of an AE began from the time that the patient provided informed consent through and including 30 calendar days after the last administration of BVD-523 (or at the time when a patient begins a new anti-cancer therapy). Anticipated fluctuations of preexisting conditions, including the disease under study that did not represent a clinically significant exacerbation or worsening, did not need to be considered AEs. AEs were collected/assessed at each study visit.
Description: A TEAE is any AE temporally assoc. with the use of BVD-523 related or not. If the onset of an AE was missing & the AE resolution date was either after the initial BVD-523 dose date or missing, then the AE was considered TE. A patient who reported multiple AEs that map to a common PT/SOC was counted only once for that PT/SOC at the highest severity reported & at the greatest relationship to study drug. AEs were assessed for all participants in Part 2 combined.
Groups:
- Cohort-expansion: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
Arm/Group | Dose-escalation 10mg b.i.d. Cohort | Dose-escalation 20mg b.i.d. Cohort | Dose-escalation 40mg b.i.d. Cohort | Dose-escalation 75mg b.i.d. Cohort | Dose-escalation 150mg b.i.d. Cohort | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Dose-escalation 900mg b.i.d. Cohort | Cohort-expansion
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/4 | 0/7 | 0/4 | 0/7 | 3/108
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/1 | 1/1 | 1/1 | 2/4 | 2/7 | 1/4 | 5/7 | 57/108
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 4/4 | 7/7 | 4/4 | 7/7 | 107/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation 10mg b.i.d. Cohort (N=1) | Dose-escalation 20mg b.i.d. Cohort (N=1) | Dose-escalation 40mg b.i.d. Cohort (N=1) | Dose-escalation 75mg b.i.d. Cohort (N=1) | Dose-escalation 150mg b.i.d. Cohort (N=1) | Dose-escalation 300mg b.i.d. Cohort (N=4) | Dose-escalation 600mg b.i.d. Cohort (N=7) | Dose-escalation 750mg b.i.d. Cohort (N=4) | Dose-escalation 900mg b.i.d. Cohort (N=7) | Cohort-expansion (N=108)
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
DISEASE PROGRESSION (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 9
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
DEATH (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FUNGAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
STRIDOR (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
FACTOR VIII INHIBITION (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
CARDIAC ARREST (Cardiac disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERICARDIAL EFFUSION (Congenital, familial and genetic disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
OVERDOSE (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — TOXICITY TO VARIOUS AGENTS
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
THROMBOSIS (Vascular disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
HYPOVOLAEMIC SHOCK (Vascular disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONVULSION (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ATAXIA (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEMIPARESIS (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PETIT MAL EPILEPSY (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GALLBLADDER OBSTRUCTION (Hepatobiliary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
HAEMATURIA (Renal and urinary disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OPTIC NERVE DISORDER (Eye disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RETINAL VEIN OCCLUSION (Eye disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIPASE INCREASED (Investigations) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIAC NEOPLASM UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DELIRIUM (Psychiatric disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ESCHERICHIA BACTERAEMIA (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UROSEPSIS (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation 10mg b.i.d. Cohort (N=1) | Dose-escalation 20mg b.i.d. Cohort (N=1) | Dose-escalation 40mg b.i.d. Cohort (N=1) | Dose-escalation 75mg b.i.d. Cohort (N=1) | Dose-escalation 150mg b.i.d. Cohort (N=1) | Dose-escalation 300mg b.i.d. Cohort (N=4) | Dose-escalation 600mg b.i.d. Cohort (N=7) | Dose-escalation 750mg b.i.d. Cohort (N=4) | Dose-escalation 900mg b.i.d. Cohort (N=7) | Cohort-expansion (N=108)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 21
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7
VISUAL IMPAIRMENT (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 10
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 12
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 25
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 3 | 6 | 59
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 9
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 6 | 49
ORAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 5 | 31
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 5
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
FATIGUE (General disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 5 | 1 | 7 | 54
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 28
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7
PYREXIA (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 20
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 8
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 13
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 11
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 5 | 38
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 19
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 10
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 8
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
DIZZINESS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 16
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 10
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 10
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 20
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 7
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 11
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3 | 36
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 18
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 31
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 26
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 11
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 5
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 31
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
PAINFUL DEFAECATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PERITONEAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HIRSUTISM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MACULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAIL BED DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NAIL GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DISEASE PROGRESSION (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 9
APPLICATION SITE RASH (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
THIRST (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
KIDNEY INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NAIL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ONYCHOMYCOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BODY TEMPERATURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OCCULT BLOOD POSITIVE (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
PROTEIN TOTAL DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ATAXIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
TENSION HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
HOT FLUSH (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
ABNORMAL SENSATION IN EYE (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHALAZION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHORIORETINOPATHY (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EYE DISCHARGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
MYDRIASIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PHOTOPHOBIA (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
EYE CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LIP INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
CONDUCTION DISORDER (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
VULVOVAGINAL ERYTHEMA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SINUS OPERATION (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT01781429/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT01781429/SAP_001.pdf